CLINICAL TRIAL: NCT04744571
Title: Safety and Efficacy of Drug-Coated Balloon Angioplasty for the Treatment of Chronic Total Occlusions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiantao Song, MD, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCB at CTO
Record Dates: First submitted 2021-02-01; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease; Coronary Occlusion; Percutaneous Coronary Intervention; Chronic Total Occlusion of Coronary Artery; Drug-Eluting Stents
Keywords: Chronic Total Occlusion; drug-coated balloon; balloon angioplasty; drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Coronary Occlusion | interventions — Aspirin; Metoprolol; Atorvastatin; Rosuvastatin Calcium; Clopidogrel; Ticagrelor; Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB group (Experimental): Patients treated with Drug-Coated Balloon Angioplasty after revascularization of Chronic Total Occlusions
  Interventions: Drug: aspirin, betaloc, atorvastatin, rosuvastatin, clopidogrel, ticagrelor; Device: coronary wires. or coronary balloons; Other: drug-coated balloon
- DES group (Active Comparator): Patients treated with Drug eluting stents Angioplasty after revascularization of Chronic Total Occlusions
  Interventions: Drug: aspirin, betaloc, atorvastatin, rosuvastatin, clopidogrel, ticagrelor; Device: coronary wires. or coronary balloons; Device: drug-eluting stent

INTERVENTIONS:
Drug: aspirin, betaloc, atorvastatin, rosuvastatin, clopidogrel, ticagrelor — Optimal medical therapy includes dual antiplatelet therapy and statins (aspirin, clopidogrel, ticagrelor, atorvastatin, rosuvastatin, betaloc). And optimal medical therapy should include adequate ventricular rate- limiting medication (i.e. Beta- blocker or rate-limiting calcium antagonist) where appropriate. Anti- anginal therapy should be used if the patients have symptom.
  Other Names: Optimal medical therapy
Device: coronary wires. or coronary balloons — all species of coronary wires, or plain balloons
Other: drug-coated balloon — Drug-coated balloon including all sizes and all brands
  Arms: DCB group
Device: drug-eluting stent — Drug-eluting stent including all sizes and all brands
  Arms: DES group

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of drug-coated balloon angioplasty for the treatment of chronic total occlusions patients with chronic total occlusion (CTO) lesion.

DETAILED DESCRIPTION:
Recruited CTO patients will be divided into two groups: those undergoing PCI of drug-coated balloon (DCB group), and those undergoing PCI of drug eluting stent implantation (DES group). The primary outcome assessed will be the late lumen loss evaluation at a 12-month of follow-up appointment. Secondary outcomes include occurrence of major cardiac events (MACEs), myocardial viability, operate success, quality of life changes which will be compared to a baseline measurement.

ELIGIBILITY:
Inclusion Criteria

* Patients between 18 and 80 years of age
* Must comply all the evaluations and follow-up protocols
* Clinical diagnosis of CTO detected using coronary angiography (at least one other major vessel should have exhibited no less than 75% stenosis)
* Patients should present with left ventricular ejection fraction (LVEF) above 35% determined using transthoracic echocardiography
* CTO located in an epicardial coronary artery with a reference diameter of ≥ 2.5 mm

Exclusion Criteria

* Patients have suffered from acute myocardial infarction within the previous 3 months
* Lesion located in the left main artery (stenosis ≥50%)
* Clinical diagnosis of rheumatic valvular disease
* Clinical diagnosis of severe arrhythmia
* With history of revascularization within the CTO artery
* Lesions unsuitable for PCI
* Severely abnormal hematopoietic systems, such as platelet counts <100 x 109/L or > 700 x 109/ L and white blood cell counts < 3 x 109/L
* Patients with active bleeding or bleeding tendencies (active ulcers, short-term ischemic stroke, history of hemorrhagic stroke, intracranial space occupying lesions, recent craniocerebral trauma, and other bleeding or bleeding tendency)
* Patients with severe coexisting condition including: severe renal function dysfunction [Glomerular filtration rate (GFR) less than 60 ml/min • 1.73 m2), severe hepatic dysfunction [glutamic-pyruvic transaminase (ALT) or glutamic-oxal acetic transaminase (ALT) elevated more than three times that of the upper limit of the normal reference], severe heart failure (NYHA classification III-IV), acute infectious diseases and immune disorders, tumors, surgery within 3 months, a life expectancy less than 12 months, pregnancy or planning to become pregnant, history of allergy or adverse reactions to aspirin, clopidogrel, ticagrelor, stains, contrast material, anticoagulant, or stents
* Patients cannot tolerate dual antiplatelet treatment (DAPT)
* Patients are unable to communicate due to cognitive impairment, auditory or visual impairment
* Patients are participating in another trial for medication or an apparatus and in which the main endpoint has not been reached, or plan to participate in a clinical trial within 12 months of the intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the difference in minimal lumen diameter (MLD) between two groups | 12 months
  Measured by Intravascular ultrasound (IVUS) or optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Comparison of the incidence of major adverse cardiac events（MACEs） between two groups | 12 months
  all-cause mortality, cardiac death, a first or recurrent, non-fatal, acute myocardial infarction, target lesion revascularization (PCI or CABG), stroke, heart failure and cardiac rehospitalization
Comparison of myocardial viability (late gadolinium enhancement, LGE) in the territory supplied by the CTO artery between two groups evaluated via cardiovascular magnetic resonance (CMR) | 12 months
  Myocardial viability in the territory supplied by the CTO artery by comparison of late gadolinium enhancement between two groups.

OTHER OUTCOMES:
Comparison of the incidence of adverse cardiac events between two groups in the perioperative period | 7 days before and after procedure
  Outcome measures including acute coronary artery occlusion, acute vascular perforation, acute stent thrombosis, acute myocardial infarction, and cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: xiantao song, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Department of Cardiology, Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided